CLINICAL TRIAL: NCT01045096
Title: A Phase 1, Randomized, Open-Label, Parallel Design, Multicenter Study to Evaluate the Pharmacokinetics and Safety of Dexlansoprazole Delayed Release Capsules in Pediatric Subjects Ages 1 to 11 Years Old With Symptomatic Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of Dexlansoprazole in Pediatric Subjects With Symptomatic Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: T-P107-174; U1111-1112-1684 (Registry Identifier: WHO)
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Erosive Esophagitis; Pharmacokinetics; Pediatrics; Drug Therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexlansoprazole 15 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole
- Dexlansoprazole 30 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole
- Dexlansoprazole 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole 15 mg, delayed release capsules, orally, once daily for up to 7 days.
  Other Names: Kapidex; TAK-390MR; Dexilant
  Arms: Dexlansoprazole 15 mg QD
Drug: Dexlansoprazole — Dexlansoprazole 30 mg, delayed release capsules, orally, once daily for up to 7 days
  Other Names: Kapidex; TAK-390MR; Dexilant
  Arms: Dexlansoprazole 30 mg QD
Drug: Dexlansoprazole — Dexlansoprazole 60 mg, delayed release capsules, orally, once daily for up to 7 days
  Other Names: Kapidex; TAK-390MR; Dexilant
  Arms: Dexlansoprazole 60 mg QD

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of dexlansoprazole, once daily (QD), in pediatric subjects with symptomatic Gastroesophageal Reflux Disease.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease (GERD) is a condition of several causes resulting in the backward flow of gastric contents into the esophagus through the lower esophageal sphincter. The prevalence of GERD in the pediatric population is increasingly becoming recognized and documented. It is a disease that may persist through adulthood, with symptoms in older children and adolescents similar to those seen in adults.

Younger children generally present with extra-esophageal manifestations, regurgitation, and epigastric pain, while older children and adolescents typically present with adult-type GERD symptoms of heartburn and regurgitation. Treatment for GERD is aimed at improving symptoms and healing esophageal inflammation.

Takeda Global Research & Development Center, Inc. (TGRD) developed dexlansoprazole delayed release capsules as a new therapy for treating acid related disorders including symptomatic non-erosive GERD, healing of erosive esophagitis (EE) and maintenance of healed EE.

Dexlansoprazole delayed release capsules have not been studied in subjects younger than 12 years of age. This study is designed to evaluate the safety of dexlansoprazole delayed release capsules in the pediatric population (1 to 11 years old) and to determine if the PK profile of dexlansoprazole in subjects 1 to 11 years of age is similar to that in adults given a similar dose.

Subjects who satisfy the screening evaluation and Inclusion/Exclusion Criteria may be enrolled in the study. Eligible subjects will be assigned to one of three treatment groups. Attempts will be made to enroll an equal number of male and female subjects in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body weight within the 5th through 95th percentile by age, inclusive, as determined by the National Center for Health Statistics .
* Females of childbearing potential must not be nursing, must have a negative serum pregnancy test at the Screening Visit and on Day -1, and if sexually active agree to routinely use adequate contraception from Screening and throughout the duration of the study.
* Subjects who take prescription or non-prescription proton pump inhibitors (PPI), histamine receptor antagonists (except cimetidine), sucralfate, or antacids on a regular or as required basis must agree to discontinue usage on Day -1 and agree to discontinue use throughout the study.
* Must have a history of GERD symptoms for at least 2 months prior to Screening or is currently symptomatic, as determined by the investigator.
* Must be able to swallow study drug capsule or must be able to ingest study drug granules sprinkled on 1 tablespoon of applesauce.

Exclusion Criteria:

* Has evidence of current cardiovascular, central nervous system, pulmonary, endocrine disease, hepatic, hematopoietic, renal, or metabolic dysfunction, serious allergy, asthma, or allergic skin rash.
* Has a known hypersensitivity to any PPI or any component of the formulation of dexlansoprazole capsules.
* Is taking any other prescription (except birth control) or nonprescription medication (including cimetidine), vitamins, or dietary supplements within 10 days prior to Day 1, or has taken herbal over-the-counter medications within 28 days prior to Day 1.
* Has a positive test result for hepatitis B surface antigen or hepatitis C virus antibody.
* Has donated or lost greater than 10% of the total blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
* Has a history of alcohol abuse or illegal drug use or drug abuse in the past, or tests positive for alcohol or drugs of abuse at the initial Screening Visit or Day -1 or is unwilling to agree to abstain from alcohol and drugs throughout the study.
* Has used a product containing nicotine within 90 days prior to the first dose of study drug or has a positive cotinine screen at the initial Screening Visit or Day -1 or is unwilling to agree to abstain throughout the study.
* Is determined to be a Cytochrome P450 2C19 poor metabolizer (ie, genotyped homozygous non-wild-type).

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (4):
- United States (4):
  - Anaheim, California
  - Miami Garden, Florida
  - Kansas City, Missouri
  - Cincinnati, Ohio

REFERENCES:
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 3 investigative sites in the United States from 04 March 2010 to 09 February 2011.
Pre-assignment Details: 36 participants with gastroesophageal reflux disease were assigned to 1 of 3 once daily (QD) treatment regimens (15 mg, 30 mg or 60 mg dexlansoprazole) based on baseline body weight.
Groups:
- Dexlansoprazole 15 mg QD: Dexlansoprazole 15 mg, delayed release capsules, orally, once daily for up to 7 days.
- Dexlansoprazole 30 mg QD: Dexlansoprazole 30 mg, delayed release capsules, orally, once daily for up to 7 days
- Dexlansoprazole 60 mg QD: Dexlansoprazole 60 mg, delayed release capsules, orally, once daily for up to 7 days
Period: Overall Study
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Started | 12 | 12 | 12
Pharmacokinetic Set | 9 (All patients with at least one estimable PK parameter for dexlansoprazole on Day 7.) | 11 | 11
Completed | 9 | 12 | 12
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 3.3 (1.97) | 7.8 (2.89) | 10.2 (0.72) | 7.1 (3.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 12
  Male | 7 | 10 | 7 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 6 | 8 | 8 | 22
  Non-Hispanic or Latino | 6 | 4 | 4 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2 | 0 | 0 | 2
  White | 8 | 12 | 12 | 32
  Multiracial | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36
Mean height [Mean (Standard Deviation); unit: cm] — Height for one patient in the Dexlansoprazole 15 mg group was incorrectly reported (as 38 cm instead of 96.52 cm) and is included in the mean height reported here. The mean height excluding this patient is 97.45 cm.
  cm | 92.5 (24.16) | 131.9 (18.80) | 146.3 (8.73) | 123.6 (29.17)
Overall Mean Weight [Mean (Standard Deviation); unit: kg] | 15.7 (5.43) | 29.7 (11.86) | 41.0 (8.50) | 28.8 (13.64)
Number of Participants per Weight Group [Number; unit: participants]
  8.6 kg - < 12.7 kg | 5 | 0 | 0 | 5
  12.7 kg - < 25.4 kg | 7 | 6 | 0 | 13
  ≥ 25.4 kg | 0 | 6 | 12 | 18
Mean Weight per Weight Group [Mean (Standard Deviation); unit: kg]
  8.6 kg - < 12.7 kg | 11.1 (1.05) | NA (NA) — There were no participants in this group | NA (NA) — There were no participants in this group | 11.1 (1.05)
  12.7 kg - < 25.4 kg | 19.0 (4.76) | 20.3 (3.67) | NA (NA) — There were no participants in this group | 19.6 (4.17)
  ≥ 25.4 kg | NA (NA) — There were no participants in this group | 39.1 (9.19) | 41.0 (8.50) | 40.3 (8.51)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Height for one patient in the Dexlansoprazole 15 mg group was incorrectly reported (as 38 cm instead of 96.52 cm) and is included in the mean BMI reported here. The mean BMI excluding this patient is 16.52 kg/m^2.
  kg/m^2 | 22.3 (20.08) | 16.4 (3.09) | 19.0 (2.56) | 19.2 (11.73)

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach the Peak Plasma Concentration (Tmax)
Description: Time to reach the maximum plasma concentration (Cmax) of Dexlansoprazole, equal to time (hours) to Cmax, as observed on Day 7. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic (PK) set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 9 | 11 | 11
hours | 4.4 (3.18) | 4.1 (2.34) | 4.1 (3.59)
Statistical Analysis 1: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 30 mg QD vs Dexlansoprazole 60 mg QD; Sample size of 12 participants per dose group, along with the intense PK sampling in each regimen was needed for characterization of the PK profile. An analysis of variance with covariates (ANCOVA) model with weight as a covariate and regimen as a factor were fitted to Tmax. Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; p = 0.809, ANCOVA

2. Other Pre Specified Outcome: Dose-normalized Peak Plasma Concentration (Cmax/Dose)
Description: Maximum observed plasma concentration (the peak plasma concentration of a drug after administration), normalized by dose. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 9 | 11 | 11
ng/mL/mg | 37.3 (15.02) | 33.5 (24.94) | 16.1 (8.65)
Statistical Analysis 1: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 30 mg QD; Sample size of 12 participants per dose group, along with the intense PK sampling in each regimen was needed for characterization of the PK profile. An ANCOVA model with weight as a covariate and regimen as a factor were fitted to dose-normalized Cmax. Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.20, 90% CI 2-sided [0.660 to 2.183]
Statistical Analysis 2: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 60 mg QD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA; Dose proportionality Point Estimate = 1.06, 90% CI 2-sided [0.463 to 2.427]
Statistical Analysis 3: Comparison: Dexlansoprazole 30 mg QD vs Dexlansoprazole 60 mg QD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 0.88, 90% CI 2-sided [0.493 to 1.579]

3. Other Pre Specified Outcome: Dose-normalized Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration (AUC(0-tlqc)/Dose)
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (tlqc), calculated using the linear trapezoidal rule, and normalized by dose. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 9 | 11 | 11
ng*hr/mL/mg | 128 (42.1) | 96 (55.6) | 62 (46.6)
Statistical Analysis 1: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 30 mg QD; Sample size of 12 participants per dose group, along with the intense PK sampling in each regimen was needed for characterization of the PK profile. An ANCOVA model with weight as a covariate and regimen as a factor were fitted to dose-normalized AUC[0-tlqc]. Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.13, 90% CI 2-sided [0.693 to 1.848]
Statistical Analysis 2: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 60 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.15, 90% CI 2-sided [0.584 to 2.276]
Statistical Analysis 3: Comparison: Dexlansoprazole 30 mg QD vs Dexlansoprazole 60 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.02, 90% CI 2-sided [0.632 to 1.642]

4. Other Pre Specified Outcome: Dose-normalized Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to 24 Hours Post-dose (AUC(0-24)/Dose)
Description: AUC(0-24) is measure of area under the curve over the dosing interval (tau), where tau is the length of the dosing interval (24 hours), calculated using the linear trapezoidal rule and normalized by dose. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 6 | 8 | 6
ng*hr/mL/mg | 143.2 (37.58) | 87.6 (46.11) | 55.5 (31.39)
Statistical Analysis 1: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 30 mg QD; Sample size of 12 participants per dose group, along with the intense PK sampling in each regimen was needed for characterization of the PK profile. An ANCOVA model with weight as a covariate and regimen as a factor were fitted to dose-normalized AUC[0-24]. Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.06, 90% CI 2-sided [0.692 to 1.636]
Statistical Analysis 2: Comparison: Dexlansoprazole 15 mg QD vs Dexlansoprazole 60 mg QD; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.26, 90% CI 2-sided [0.691 to 2.314]
Statistical Analysis 3: Comparison: Dexlansoprazole 30 mg QD vs Dexlansoprazole 60 mg QD; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; ANCOVA; Dose Proportionality Point Estimate = 1.19, 95% CI 2-sided [0.777 to 1.817]

5. Primary Outcome: The Peak Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 9 | 11 | 11
ng/mL | 559 (225.3) | 1005 (748.1) | 964 (519.0)

6. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration (AUC(0-tlqc))
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (tlqc), calculated using the linear trapezoidal rule. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 9 | 11 | 11
ng*hr/mL | 1914 (631.8) | 2892 (1668.6) | 3747 (2795.6)

7. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to 24 Hours Post-dose (AUC(0-24))
Description: AUC(0-24) is measure of area under the curve over the dosing interval (tau), where tau is the length of the dosing interval (24 hours), calculated using the linear trapezoidal rule. Pharmacokinetic parameters were derived using noncompartmental methods from the plasma concentrations of dexlansoprazole.
Time Frame: Day 7 after 7 days of dosing with dexlansoprazole delayed release capsules.
Population: Pharmacokinetic set included all participants with at least one estimable PK parameter for dexlansoprazole on Day 7.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Number analyzed (Participants) | 6 | 8 | 6
ng*hr/mL | 2149 (563.7) | 2628 (1383.2) | 3330 (1883.3)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events with an onset that occurred after receiving study drug and within 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole 15 mg QD | Dexlansoprazole 30 mg QD | Dexlansoprazole 60 mg QD
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 5/12 | 2/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 15 mg QD (N=12) | Dexlansoprazole 30 mg QD (N=12) | Dexlansoprazole 60 mg QD (N=12)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 15 mg QD (N=12) | Dexlansoprazole 30 mg QD (N=12) | Dexlansoprazole 60 mg QD (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of it's obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.